CLINICAL TRIAL: NCT06708507
Title: A Prospective Study on the Correlation Between Tissue-resident Immune Cell Subsets and Graft-versus-host Disease Following Hematopoietic Stem Cell Transplantation.
Brief Title: Tissue-resident Immune Cell Subsets in aGVHD
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2024-084
Record Dates: First submitted 2024-11-17; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Acute Graft-versus-Host Disease; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 100 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Grade 3-4 aGVHD patients
- Grade 1-2 aGVHD patients

SUMMARY:
This is a prospective study investigating the role of tissue-resident immune cell subsets in the occurrence and progression of graft-versus-host disease following hematopoietic stem cell transplantation. Approximately 40 subjects(including 20 grade 3-4 aGVHD patients and 20 grade 1-2 aGVHD patients ).

DETAILED DESCRIPTION:
This study was a single-center, observational, prospective cohort study. The study lasted for 3 months, from 2024.11 to 2025.02.It is planned to enroll 40 subjects, divided into 20 grade 3-4 aGVHD patients and 20 grade 1-2 aGVHD patients. No randomization or any protocol-driven treatment will be performed or provided to subjects during the course of the study. Treatment decisions and selection of treatment options are left to the discretion of the treating physician, if clinically appropriate. All recipients will be followed for aGVHD evaluation,overall survival(OS) ,disease-free survival (DFS). aGVHD were graded according to published guidelines. All recipients will be monitored every month until the study is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form;
2. Age 16-65 years old
3. Clinically diagnosed with GVHD for the first time/receiving GVHD treatment.

Exclusion Criteria:

1. Have a history of other tumors
2. With poor compliance or mental disorders
3. Infected with HIV and HCV
4. With uncontrolled HBV infection
5. With other autoimmune diseases
6. Those who are judged by the researcher to be unsuitable to participate in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients develop acute graft-versus-disease after hematopoietic stem cell transplantation.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Association between tissue-resident Immune cell subsets in organ and acute graft-vs-host disease (aGVHD) outcomes. | 100days
  Measure the number/proportion of resident T,B and macrophage cell subsets in the main organ of aGVHD(skin,intestine and liver).

SECONDARY OUTCOMES:
Association between tissue-resident Immune cell subsets in organ and overall survival(OS). | 100days
  Measure the number/proportion of resident T,B and macrophage cell subsets in the main organ of aGVHD(skin,intestine and liver).
Association between tissue-resident Immune cell subsets in organ and disease-free survival (DFS) | 100days
  Measure the number/proportion of resident T,B and macrophage cell subsets in the main organ of aGVHD(skin,intestine and liver).

CONTACTS AND LOCATIONS:
Overall Officials: Hua Jin, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No